CLINICAL TRIAL: NCT02430025
Title: Fujian Province Cardiovascular Diseases Study
Acronym: FJCVD
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Fujian Provincial Hospital (Other)
Collaborators: Peking University (Other)
Responsible Party: Principal Investigator, Guo Yansong, Director of the cardiology department, Fujian Provincial Hospital
Other Study IDs: FJPH20150101
Record Dates: First submitted 2015-04-23; First posted 2015-04-29 (Estimated); Last update posted 2015-04-29 (Estimated); Status verified 2015-04

CONDITIONS: Cardiovascular Diseases
Keywords: Cardiovascular Diseases; Vascular Diseases; Acute Coronary Syndrome; Chest Pain; Heart Diseases; Myocardial Ischemia; Pathologic Processes
MeSH Terms: conditions — Cardiovascular Diseases; Vascular Diseases; Acute Coronary Syndrome; Chest Pain; Heart Diseases; Myocardial Ischemia; Pathologic Processes

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Approximately 30 mls of blood will be dispensed as follows :
  3 x 10 mls EDTA Tube (Blood was collected from overnight-fasted subjects into ice-cold tubes containing EDTA) (6 mmol/L final concentration).
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (4):
- control subjects: people had no clinical history of cardiovascular diseases,no family history of premature cardiovascular diseases.
- coronary atherosclerosis: Subjects with CAD also had at least one <50% stenotic lesion on coronary angiography.
- stable coronary artery disease: Subjects with stable CAD had clinically established atherosclerotic vascular disease but had been stable for ≥3 months.
- acute coronary syndrome: Subjects with CAD also had at least one ≥50% stenotic lesion on coronary angiography or a history of myocardial infarction, percutaneous coronary intervention, or coronary artery bypass grafting. All subjects with ACS exhibited acute ECG changes consistent with myocardial ischemia or elevated troponin levels. ACS was confirmed with urgent coronary angiography; all subjects had at least one ≥50% stenotic lesion with ruptured plaque or thrombus.

SUMMARY:
This proposal delineates a research plan to collect blood from the patients with cardiovascular diseases for the purpose of establishing a molecular biological bank registry. The Fujian provincial hospital will enroll 8,000 patients.The blood collected will be processed to create a repository of molecular biological plasma. Along with a sample of blood collected from individual patients, a concise general medical history, demographic data, electrocardiographic data, echocardiographic data, and laboratory data will be collected. A short interview will take place after enrollment during the outpatient visit or hospital stay, or may be conducted via phone call after enrollment. All the clinical data gathered will be compiled in Fujian provincial hospital center database, and would be stored in a format where a culmination of clinical findings, i.e. representing a disease of interest, can be used to search the database to identify the blood samples of all patients with such characteristics for further study.

DETAILED DESCRIPTION:
The study is to commence on May 1st 2015 and is to be completed within 3-5 years. The targeted number of patients to be enrolled is 8,000. All patients have the history of cardiovascular diseases, will be eligible to be enrolled. Patients inclusion criteria are as follows, once informed consent is obtained:

1. Males or females at least 18 years old.
2. Patient has not been previously enrolled in the molecular biological bank registry of the Fujian provincial hospital.
3. Patient able to give informed consent.
4. Any patient with history of cardiovascular diseases (If a subject reports history of cardiovascular diseases at another facility, outside records will be obtained to confirm the diagnosis.

ELIGIBILITY:
Inclusion Criteria:

* 18-80 year old males and non-child-bearing period females.
* Clinical diagnosed with acute coronary syndrome including NSTE-ACS ,MI and STEMI.
* Patients with STEMI((ST segment elevation myocardial infarction) and NSTEMI(non-ST segment elevation myocardial infarction) will be recruited within 48 hours of symptom onset.
* Patients with cerebrovascular disease was made or confirmed by a board-certified neurologist with fellowship training in cerebrovascular disease and confirmed by standard diagnostic techniques such as head CT, MRI, MR angiography, CT angiography, carotid ultrasound, etc.
* Sign the ICF(inform consent form)

Exclusion Criteria:

* child-bearing women
* hypothyroidism,
* active liver disease or dysfunction including agnogenic serum transaminase sustained elevation or higher than 3 times ULN(upper limit of normal)
* severe anemia (hemoglobin,hematocrit < 28%)
* A history of psychiatric disorders
* A history of jejunoileal bypass or gastric bypass surgery
* Currently take steroids therapy
* Diagnosed with malignant within 5 years
* Severe renal function damage (creatinine clearance rate<30 ml/min)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The control subjects had no clinical history of cardiovascular diseases, no family history of premature cardiovascular diseases.Subjects had all arteries<50% stenotic lesion on cardiocerebral vascular angiography. Subjects with stable CAD had clinically established atherosclerotic vascular disease but had been stable for ≥3 months. Subjects with CAD also had at least one ≥50% stenotic lesion on coronary angiography or a history of myocardial infarction, percutaneous coronary intervention, or coronary artery bypass grafting. ACS was confirmed with urgent coronary angiography; all subjects had at least one ≥50% stenotic lesion with ruptured plaque or thrombus.
Sampling Method: Probability Sample
Enrollment: 8000 (Estimated)
Dates: Start 2015-06; Primary Completion 2020-05 (Estimated); Study Completion 2020-05 (Estimated)

PRIMARY OUTCOMES:
To further find some unknown small Metabolic molecules by mass spectrometry | 3-5 years

CONTACTS AND LOCATIONS:
Overall Officials: yan so Guo, doctorate, Study Director — Fujian Provincial Hospital

REFERENCES:
- [Derived] Chen X, Guo Y, Lai L, Zhang S, Li Z. Intracoronary and peripheral blood levels of TNF-like Cytokine 1A (TL1A) in patients with acute coronary syndrome. Medicine (Baltimore). 2020 May 29;99(22):e20305. doi: 10.1097/MD.0000000000020305. PMID 32481400